CLINICAL TRIAL: NCT07287124
Title: A Pivotal, Pre-market, Prospective, Interventional, Multi-centre Study to Evaluate Clinical Benefit, Performance, and Safety of the TI1132 Implant in an Adult Population With Sensorineural Hearing Loss
Brief Title: A Pivotal Study to Evaluate the Clinical Benefit, Performance and Safety of a Totally Implantable Cochlear Implant (TICI) System in Adults
Acronym: ELEVATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5828
Record Dates: First submitted 2025-12-11; First posted 2025-12-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss, Bilateral Sensorineural
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Totally Implantable Cochlear Implant System (Experimental): Participants will be implanted with the TI1132 implant
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — Totally Implantable Cochlear Implant System

SUMMARY:
This pivotal study examines the clinical efficacy and safety of an investigational totally implantable cochlear implant (TICI) system. The system includes a microphone placed under the skin to detect speech and sound from the environment, providing the option to hear without any visible external parts. This study will involve adults with sensorineural hearing loss, a type of hearing loss caused by damage to the inner ear or auditory nerve (the nerve that carries sound signals from the ear to the brain). Participants will complete hearing tests and questionnaires to evaluate how well the system works and how it affects their daily life.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and older at time of consent.
* Clinically established sensorineural hearing loss (SNHL) defined by a four frequency (500, 1000, 2000, 4000 Hz) pure-tone average unaided threshold (PTA4) of ≥70 dB HL in the ear to be implanted.
* Compromised functional hearing in the aided condition defined as ≤40% correct on a word recognition test in the ear to be implanted.
* Clinically established SNHL defined by a four-frequency (500, 1000, 2000 & 4000 Hz) pure-tone average unaided threshold (PTA4) of ≥30 dB HL in the contralateral ear.
* Candidate is a fluent speaker in the language used to assess speech perception performance as determined by the investigator.
* Direct access to a compatible Smart Phone.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Prior cochlear implantation, in either ear, or medical plan for cochlear implantation during the clinical investigation, contralateral to the ear to be implanted.
* Candidates with single-sided deafness as determined by the investigator.
* Intra-axial (within-the-brain) lesions or deafness due to lesions of the acoustic nerve affecting the ear to be implanted.
* Middle ear infection (including acute otitis media, chronic otitis media, suppurative otitis media, or serous drainage) in the ear to be implanted either at the time of surgery or within 3 months prior to enrolment.
* Presence of a tympanic membrane perforation or a history of otologic surgery within 3 months prior to enrolment, in the ear to be implanted.
* Previously reported diagnosis of auditory neuropathy, in the ear to be implanted.
* Ossification, malformation or any other cochlear anomaly, such as common cavity, that might prevent complete insertion of the electrode array, in the ear to be implanted.
* Current cerebrospinal fluid (CSF) shunts or drains, existing perilymph fistula, skull fracture or CSF leaks.
* Severe, or poorer, bilateral sensorineural hearing loss prior to 5 years of age, as reported by the participant.
* Severe, or poorer, sensorineural hearing loss for more than 20 years, as reported by the participant, in the ear to be implanted.
* Medical or psychological conditions that contraindicate general anaesthesia, surgery, or participation in the clinical investigation as determined by the investigator.
* Pre-existing skin condition that could jeopardize wound healing as judged by the investigator e.g., psoriasis, dermatitis, use of corticosteroids, uncontrolled diabetes.
* Unrealistic expectations on the part of the participant, regarding the possible benefits, risks, and limitations inherent to the surgical procedure(s) and prosthetic devices, as determined by the Investigator.
* Additional disabilities that may affect the participant's participation or safety during the clinical investigation.
* Unable or unwilling to comply with all requirements of the clinical investigation, as determined by the investigator.
* Pregnant or breastfeeding women.
* Investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as spouse, parent, child or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of the investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless Cochlear sponsored and determined by Investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Speech recognition performance in quiet | Preimplantation to 6-months post-activation
  Percent correct scores in word recognition score from pre-implantation to post-implantation.
Incidence of adverse events and device deficiencies | Implantation to 6- and 12-months post-activation
  Frequency and severity of device and procedure-related adverse events, including device deficiencies.

SECONDARY OUTCOMES:
Speech, Spatial and Qualities of Hearing questionnaire (SSQ-12) | Preimplantation to 6- and 12-months post-activation
  Speech, Spatial, and Qualities of Hearing Scale global score (SSQ-12). Scores range from 0 to 10, where higher scores indicate greater ability (less hearing disability).
Speech recognition performance in noise | Preimplantation to 6- and 12-months post-activation
  Percent correct sentence score from preimplantation to 6- and 12-months post-activation.
Speech recognition performance in quiet | Preimplantation to 12-months post-activation
  Percent correct word recognition score in quiet from pre-implantation to post-implantation.
Cochlear Implant Quality of Life Profile (CIQOL-35) | Preimplantation to 6- and 12-months post-activation
  Cochlear implant hearing related quality of life score (CIQOL-35). Scored for six health domains (communication, emotional, entertainment, environment, listening effort, and social) each scaled from 0 to 100, where a higher score indicates better health.
Health Utilities Index (HUI 2/3) | Preimplantation to 6- and 12-months post-activation
  Health Utilities Index (HUI 2/3) global score. Scores range from -0.36 to 1.00, where a negative score represents a state "worse than dead" and a top score of 1.00 is "perfect health".
Living with Cochlear Implants Questionnaire (LivCI) | Preimplantation to 6- and 12-months post-activation
  Living with Cochlear Implants Questionnaire (LivCI) evaluates the impact of a hearing device on four domains, Participation (range 0 to 12), Psychosocial & Wellbeing (range 0 to 21), Stigma (range 0 to 15) and Management & Aesthetics (range 0 to 18), where a higher domain score indicates positive patient report.
Patient Satisfaction Survey | From 6 to 12 months post-activation
  Device satisfaction rating score. Scores range from 1 to 5, where a higher score indicates greater patient satisfaction with the TICI system.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Buchman, Principal Investigator — University of Utah
Locations (11):
- United States (11):
  - Rocky Mountain Ear Center, Englewood, Colorado
  - University of Miami School of Medicine, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - Michigan Ear Institute, Novi, Michigan
  - Mayo Foundation Rochester, Rochester, Minnesota
  - Midwest Ear Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - New York University, New York, New York
  - University Hospitals Cleveland Medical Centre, Beachwood, Ohio
  - Hearts for Hearing Foundation, Oklahoma City, Oklahoma
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No